CLINICAL TRIAL: NCT04716855
Title: Evaluation of Daily Life Activities in Patients With Rotator Cuff Syndrome
Brief Title: Evaluation of Functional Status, Physical Activity and Quality of Life in Patients With Rotator Cuff Syndrome
Status: Completed | Type: Observational
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 10840098-604.01.01-E.4606.
Record Dates: First submitted 2021-01-16; First posted 2021-01-20 (Actual); Last update posted 2021-01-20 (Actual); Status verified 2015-03

CONDITIONS: Rotator Cuff Syndrome
Keywords: Pain; Physical activity; Rotator cuff syndrome; Quality of life
MeSH Terms: conditions — Pain; Motor Activity | interventions — Quality of Life

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Evaluation tests: RCS cases between the ages of 19-64 (n:40) who agreed to participate were included in the study. Pain severity (Visual Analogue Scale - VAS), range of motion (Universal Goniometer), muscle test (Manual muscle test), upper extremity functional status and disability (Quick-DASH questionnaire), physical activity level (International Physical Activity Questionnaire - UFAA) ) and quality of life (Short Form-36 - SF-36) were evaluated
  Interventions: Other: Quality of life and daily living activities assessment tests

INTERVENTIONS:
Other: Quality of life and daily living activities assessment tests

SUMMARY:
Pain is one of the most important factors affecting the quality of life. The quality of life of patients with pain and restricted shoulder movements can be affected in patients with Rotator Cuff Syndrome (RCS).

DETAILED DESCRIPTION:
The aim of our study is to examine the effect of the pain on functional status, quality of life and physical activity levels in daily life activities of RCS patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting with shoulder pain problems and diagnosed with RCS.
* Individuals between the ages of 19-64 were included in the study.

Exclusion Criteria:

* Those who have mental disability at the level of understanding the test and preventing interviews.
* Those with any chronic problems (such as cancer, kidney failure)
* Those who receive special medical treatment (steroid therapy, chemotherapy, insulin use.)
* Those who had a pregnancy status were excluded from the study.

Ages: 19 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: This study was applied patients which were diagnosed with RC syndrome the Physical Therapy and Rehabilitation Department at Istanbul Medipol Mega University Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2015-03-25; Primary Completion 2016-05-20 (Actual); Study Completion 2016-12-22 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale | 2 min
  The Visual Analog Scale (VAS) is used to convert some values that cannot be measured numerically to digital. Two end definitions of the parameter to be evaluated are written on both ends of a 100 mm line and the patient is asked to indicate where his condition is appropriate by drawing a line or by placing a point or pointing on this line. In this study, the severity of pain was questioned as 1- Night pain 2- Rest pain 3- Activity pain 4- Lift pain and it was marked separately for each situation.
The Shortened Disabilities of the Arm, Shoulder and Hand Score | 10 min
  The "Quick-DASH" (The Disabilities of the Arm, Shoulder and Hand Score) questionnaire, which is the short form of the "DASH" questionnaire, was used to determine the level of activity and engagement from the upper side. The Turkish reliability and validity study of the questionnaire was carried out by Düger et al.. Each answer is scored from 1 to 5 from good to bad; 1: no difficulty, 2: mild difficulty, 3: moderate difficulty, 4: extreme difficulty, 5: not being able to do it at all. A score between 0-100 (0 = no disability, 100 = maximum disability) is obtained from each part of the Quick-DASH questionnaire.
Short Form-36 (SF-36) | 10 min
  Short Form SF-36 was used to evaluate the quality of life. SF-36 consists of 8 sub-dimensions consisting of 36 items in which physical and mental health is evaluated. The Turkish reliability and validity study of the questionnaire was carried out by Koçyiğit et al. [21]. There are two main subsections belonging to SF-36. In the physical health components subsection are included Physical function (PF), physical role (PR), body pain (BP) and general health status (GHS) sub-dimensions. Sub-dimensions related to mental health status are stated as vitality (VT), social function (SF), emotional role (RE), and mental health (MH).
International Physical Activity Questionnaire (IPAQ) | 10 min
  It has been explained that IPAQ is a safe and valid application in determining physical activity. The Turkish reliability and validity study of the questionnaire was carried out by Ozturk.
  The questionnaire consists of 4 separate sections and includes 7 questions in total. This questionnaire includes questions about physical activity for a minimum of 10 minutes in the last 7 days.

SECONDARY OUTCOMES:
Manual Muscle Test | 10 min
  Shoulder flexion (Muscle (M)-FL), abduction (M-AB), extension (M-EX), adduction (M-AD), external rotation (M-ER) and internal rotation (M-İR) are scored by scoring between 0 and 5 in manual muscle test.
Range of Motion | 10 min
  Flexion, extension, abduction, adduction, internal rotation and external rotation range of motion were measured with a universal goniometer for the shoulder joint. The measurement values were recorded in degrees. Normal values for shoulder range of motion are 0-180º in flexion (FL) and abduction (AB), 0-45º in extension (EX) and adduction (AD), 0-90º in external rotation (ER) and 0-70º in internal rotation (IR).

CONTACTS AND LOCATIONS:
Overall Officials: Mehmet Salih Tan, Principal Investigator — Istanbul Medipol University Hospital
Locations (1):
- Istanbul Medipol University Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No